CLINICAL TRIAL: NCT02371876
Title: User Performance of the ONYX PLUS Blood Glucose Monitoring System
Brief Title: Evaluation of an Ascensia Diabetes Care ONYX PLUS Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCA-2014-005-01
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2016-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Users of the Monitoring System (Experimental): Untrained subjects with diabetes used the ONYX PLUS Investigational Blood Glucose Monitoring System.
  Interventions: Device: ONYX PLUS Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: ONYX PLUS Investigational Blood Glucose Monitoring System — Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood (and study staff tested subject fingerstick blood) using the ONYX PLUS Investigational Blood Glucose Monitoring System. All BG results were compared to reference method results obtained from subject capillary blood. Study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.

SUMMARY:
The purpose of this study was to determine if untrained subjects with diabetes can operate the Investigational ONYX PLUS Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 18 years of age and older
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or other bleeding disorder
* Pregnancy
* Physical, visual, or neurological impairments that would make the person unable to perform testing with the BGM
* Previously participated in a BG monitor study using the ONYX PLUS BGMS
* Working for a medical laboratory, hospital, or other clinical setting that involves training on or clinical use of blood glucose monitors
* Working for a competitive medical device company, or having an immediate family member who works for such a company
* A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk

The enrollment goal for the intended use population:

1. At least 70% of subjects will be younger than age 65
2. At least 20% of subjects will have type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute Inc.; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Users of the Monitoring System
Started | 134
Completed | 134
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 134
Age, Continuous [Mean (Full Range); unit: years] | 54.0 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants] — Subjects provided more than one choice for Race. Therefore, the apparent frequency total for Race was different from the number of subjects.
  participants
    American Indian or Alaska Native | 3
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 14
    White | 112
    More than one race | 3
    Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 134

OUTCOME MEASURES:

1. Primary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) and +/- 15% (>= 100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Measure: Number; unit: Percentage of BG Results
Groups:
- Users of the Monitoring System: Untrained subjects with diabetes used the ONYX PLUS Investigational Blood Glucose Monitoring System.
  ONYX PLUS Investigational Blood Glucose Monitoring System: Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick blood using the ONYX PLUS Investigational Blood Glucose Monitoring System. All BG results were compared to reference method results obtained from subject capillary blood.
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 134
Percentage of BG Results | 99.2

2. Secondary Outcome: Percent of Alternate Site Palm Blood Glucose (BG) Results Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested Alternate Site (AST) palm blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) and +/- 15% (>= 100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 126 (134-8) Blood glucose results were analyzed. Four subjects with low blood sugar did not attempt palm testing per protocol. Four subjects had low blood sugar; their palm results were not evaluable per protocol.
Measure: Number; unit: Percentage of BG Results
Groups:
- Users of the Monitoring System: Untrained subjects with diabetes used the ONYX PLUS Investigational Blood Glucose Monitoring System.
  ONYX PLUS Investigational Blood Glucose Monitoring System: Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary palm blood using the ONYX PLUS Investigational Blood Glucose Monitoring System. All BG results were compared to reference method results obtained from subject capillary blood.
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 126
Percentage of BG Results | 99.2

3. Secondary Outcome: Percent of Subject Fingerstick Blood Glucose (BG) Results Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method When Tested by Study Staff
Description: Study staff tested subject fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15mg/dL (<100mg/dL YSI capillary plasma) and +/- 15% (>= 100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Measure: Number; unit: Percentage of BG Results
Groups:
- Users of the Monitoring System: Untrained subjects with diabetes used the ONYX PLUS Investigational Blood Glucose Monitoring System.
  ONYX PLUS Investigational Blood Glucose Monitoring System: Study staff tested subject fingerstick blood using the ONYX PLUS Investigational Blood Glucose Monitoring System. All BG results were compared to reference method results obtained from subject capillary blood.
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 134
Percentage of BG Results | 99.2

4. Secondary Outcome: Percent of Venous Blood Glucose (BG) Results Within +/- 15mg/dL (<100mg/dL) and Within +/- 15% (>=100mg/dL) of Laboratory Glucose Method
Description: Study staff tested subject venous blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 15mg/dL (<100mg/dL YSI venous plasma) and +/- 15% (>= 100mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: 132 (134-2) Blood glucose results were analyzed. Venipunctures were unsuccessful for two subjects.
Measure: Number; unit: Percentage of BG Results
Groups:
- Users of the Monitoring System: Untrained subjects with diabetes used the ONYX PLUS Investigational Blood Glucose Monitoring System.
  ONYX PLUS Investigational Blood Glucose Monitoring System: Study staff tested subject venous blood using the ONYX PLUS Investigational Blood Glucose Monitoring System. BG results were compared to reference method results obtained from subject venous plasma.
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 132
Percentage of BG Results | 100

5. Secondary Outcome: Percent of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 12.5mg/dL (<100mg/dL) and Within +/- 12.5% (>=100mg/dL) of Laboratory Glucose Method
Description: Untrained subjects with diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the percent of BGMS results within +/- 12.5mg/dL (<100mg/dL YSI capillary plasma) and +/- 12.5% (>= 100mg/dL YSI capillary plasma).
Time Frame: 1 hour
Measure: Number; unit: Percentage of BG Results
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 134
Percentage of BG Results | 98.5

6. Secondary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements Regarding BGMS
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' or 'Agree' or 'Neutral' or 'Disagree' or 'Strongly Disagree'. The percent of subjects who provided responses that were 'Strongly Agree','Agree','Neutral' about each statement was calculated.
Time Frame: 1 hour
Measure: Number; unit: Percentage of Participants Who Responded
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 134
Percentage of Participants Who Responded
  I find it easy to do a blood test with this meter. | 99.2
  The meter display was easy to see and read. | 98.5
  It was easy to understand my test results. | 100
  I like the overall meter design. | 97.8
  I find the meter easy to use. | 100
  The instructions were easy to understand. | 96.3
  Instructions clearly explain how to run a test. | 97.8
  Instructions clearly explain meter error messages. | 99.2

7. Secondary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements Regarding Views/Behaviors Related to Self-Monitoring Blood Glucose
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on views and behaviors related to managing their diabetes. Subjects could respond 'Strongly Agree' or 'Agree' or 'Neutral' or 'Disagree' or 'Strongly Disagree' or 'No Answer or Not Applicable'. The percents (of subjects who responded) that were 'Strongly Agree','Agree','Neutral' about views/behaviors related to self-monitoring blood glucose were calculated.
Time Frame: 1 hour
Population: Percent (of those who responded) who 'Strongly Agree', 'Agree', 'Neutral' was calculated for each statement. Abbreviations used: 'HCP' is HealthCare Professional and 'Acc' is Accuracy
Measure: Number; unit: Percentage of Participants Who Responded
Arm/Group | Users of the Monitoring System
Number analyzed (Participants) | 134
Percentage of Participants Who Responded
  Acc:important to help me talk w my HCP. | 99.25
  Acc:important to help w self-monitor satisfaction. | 99.25
  Acc:important to help w managing my diabetes. | 100
  Acc:important to help prevent low blood sugar | 100
  Acc:important to understand food/exercise effects. | 100
  Acc:help w using results to better control diabete | 100
  Acc:important to achieve greater peace of mind. | 100
  I prefer the meter I just used to my regular meter | 86.5
  I use my meter - my care provider gave it to me. | 84.1
  I use my current meter -my insurance covers strips | 80
  I use my current meter-I think it is most accurate | 86.9

ADVERSE EVENTS:
Time Frame: Subject visits were approximately 1 hour.
Arm/Group | Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/134
Other Adverse Events (participants affected / at risk) | 4/134
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Users of the Monitoring System (N=134)
Hypoglycemia (Endocrine disorders) | 4 (4) — Subjects' hypoglycemia were resolved at the visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days